CLINICAL TRIAL: NCT06962748
Title: End-tidal Carbon Dioxide as a Non-invasive Predictor for Changes in Cardiac Output in Non-cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Adham Haggag, Dr, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: FMASU R95/2025
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Non Cardiac Surgery
Keywords: ETCO2- Cardiac output-Carotid blood flow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ETCO2 (Active Comparator): The patients EtCO2 will be recorded and the average of the reading over a time interval of 30 minutes will be recorded and correlated to the cardiac output as measured by both the carotid blood flow and the TTE
  Interventions: Diagnostic Test: ETCO2
- TTE CO (Active Comparator): a transthoracic echocardiography will be done to measure the cardiac output
  Interventions: Diagnostic Test: TTE CO measurment
- carotid blood flow (Active Comparator): The patients' Cardiac output as measured before will be correlated with the carotid blood flow after scanning the carotid artery to exclude a significant lesion as measured by the following equation and the average of a three consecutive reading will be recorded
  Interventions: Diagnostic Test: cerebral blood flow measurment

INTERVENTIONS:
Diagnostic Test: cerebral blood flow measurment — measuring CO using cerebral blood flow
  Arms: carotid blood flow
Diagnostic Test: TTE CO measurment — measuring CO using TTE
  Arms: TTE CO
Diagnostic Test: ETCO2 — measure the average ETCO2 over 30 minutes period
  Arms: ETCO2

SUMMARY:
Cardiac output (CO) is challenging to measure at the bedside. The traditional gold standard for measuring CO requires the insertion of a pulmonary artery catheter which is invasive, associated with a risk for serious complications [3],with no clinical benefits.

The cerebral blood flow (CBF) is considered to be a proportion of total cardiac output (CO). It has been stated earlier that approximately 15% of resting CO is distributed to the brain. Therefore, the flow through the CCA might serve as a surrogate parameter for CO.

DETAILED DESCRIPTION:
* Type of Study: Cross-sectional study
* Study Setting: Operating rooms at Ain Shams University Hospital
* Study Period : 6 months
* Study Population:
* Sampling Method: The study is a double blinded observational study that will be conducted at Ain Shams University hospitals on patients scheduled for Abdominal or lower limb surgeries. The patients will be randomly divided into two equal groups group D and group C Randomization will be done by computer-generated number lists and using opaque sealed envelopes.
* Sample Size: Using PASS 15 program for sample size calculation, setting confidence level at 95% and two-sided confidence interval width at 0.2, it is estimated that sample size of 105 patients will be needed to detect an expected Pearsons correlation coefficient of 0.7 between end-tidal carbon dioxide and cardiac output during surgery.
* Ethical Considerations: The study will be approved by the Research Ethics Committee of the Faculty of Medicine and conducted in accordance with the principles of the declaration of Helsinki. Written informed consent from all participants will be obtained.

Study Procedures:

After the patients consented and after the induction of the anesthesia, a transthoracic echocardiography will be done to measure the cardiac output, where the LVOT diameter is measured from the parasternal long axis view to calculate the radius of the LVOT, and the velocity time integral (VTI) is calculated from the apical five chamber and the apical three chamber view, and by applying the equation the cardiac output will be calculated CO= π* (LVOT radius)2* (LVOT VTI) *HR The patients will be monitored using electrocardiography, non-invasive blood pressure measurement and pulse oximetry (SpO2), general anesthesia will be induced using Propofol 2mg/Kg, Rocuronium 0.5mg/Kg and fentanyl 1ug/kg and the all the patients will be intubated with an endotracheal tube size 7 for female and 8 for males A warming blanket will be ensured to all the patients to maintain the core temperature at 36ْC For all the patients involved in the study. The patients' Cardiac output as measured before will be correlated with the carotid blood flow after scanning the carotid artery to exclude a significant lesion as measured by the following equation and the average of a three consecutive reading will be recorded, these will be repeated every 30 min. for the procedures.

π* (Carotid diameter )4/4* VTI *HR The carotid blood flow will be measured by applying a linear probe along the medial aspect of the sternocleidomastoid muscle above the common carotid artery, by applying pulsed wave, the pulse of the carotid artery will be traced and the VTI automatically calculated the machine. The patients EtCO2 will be recorded and the average of the reading over a time interval of 30 minutes will be recorded and correlated to the cardiac output as measured by both the carotid blood flow and the TTE .The blood pressure, heart rate will be monitored and recorded

ELIGIBILITY:
Inclusion Criteria:

* The patients age will be ranged from 18-55 years,
* ASA physical status I-II,
* General surgeries not involving the head and neck
* Orthopedic surgeries involving the lower limb
* Patients in supine posture

Exclusion Criteria:

* Those with Respiratory disease including but not limited to Pneumonia, COPD, Restrictive lung disease and ARDS
* Those with anemia.
* Patients' refusal to participate in the study.
* Thoracic surgeries.
* Morbidly obese patients.
* Significant carotid artery disease.
* Surgeries of less than 2-hour duration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
correlation of ETCO2 | during operation
  we assume that the change in the gradient of carbon dioxide release over a time in mechanically ventilated patients may be directly proportionate to the cardiac output and could reflect it.
  In the current study we will correlate the aforementioned hypothesis with the change in the cardiac output compared to the change in the carotid blood flow as revealed by the change in the cardiac output as measured by the transthoracic echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasiya, Egypt